CLINICAL TRIAL: NCT02072330
Title: A Randomized, Double-Blind, Multicenter, Phase 2/3 Study to Evaluate the Efficacy and Safety of Combined Administration of TAK-536CCB (Fix-dose Combination of Azilsartan and Amlodipine) and Hydrochlorothiazide in Comparison With TAK-536CCB or Hydrochlorothiazide Monotherapy in Patients With Grade I or II Essential Hypertension
Brief Title: Study to Evaluate the Efficacy and Safety of Combined Administration of TAK-536CCB and Hydrochlorothiazide in Patients With Grade I or II Essential Hypertension.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-536TCH/CCT-001; JapicCTI-121962 (Registry Identifier: Japic CTI)
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Grade I or II Essential Hypertension
Keywords: Hypertension, Drug therapy
MeSH Terms: conditions — Lymphoma, Follicular; Hypertension | interventions — Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- TAK-536CCB 20 mg/5 mg ＋Placebo (dual therapy) (Active Comparator): TAK-536CCB 20 mg/5 mg and Hydrochlorothiazide (HCTZ) placebo for 10 weeks
  Interventions: Drug: TAK-536CCB
- TAK-536CCB 20 mg/5 mg ＋HCTZ 6.25 mg (triple therapy) (Experimental): TAK-536CCB 20 mg/5 mg and Hydrochlorothiazide placebo (triple therapy) for the first 2 weeks of the treatment period and TAK-536CCB 20 mg/5 mg and HCTZ 6.25 mg for the remaining 8 weeks.
  Interventions: Drug: TAK-536CCB + Hydrochlorothiazide
- TAK-536CCB 20 mg/5 mg ＋HCTZ 12.5 mg (triple therapy) (Experimental): TAK-536CCB 20 mg/5 mg and Hydrochlorothiazide placebo for the first 2 weeks of the treatment period and TAK-536CCB 20 mg/5 mg and HCTZ 12.5 mg (triple therapy) for the remaining 8 weeks.
  Interventions: Drug: TAK-536CCB + Hydrochlorothiazide
- Placebo ＋HCTZ 6.25 mg (HCTZ monotherapy) (Active Comparator): TAK-536CCB placebo and Hydrochlorothiazide 6.25 mg (HCTZ monotherapy) for 10 weeks from the start of the treatment period.
  Interventions: Drug: Hydrochlorothiazide
- Placebo ＋Hydrochlorothiazide 12.5 mg (HCTZ monotherapy) (Active Comparator): TAK-536CCB placebo and Hydrochlorothiazide 12.5 mg (HCTZ monotherapy) for 10 weeks from the start of the treatment period.
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: TAK-536CCB — TAK-536CCB 20 mg/5 mg ＋Hydrochlorothiazide placebo tablets
  Other Names: Fix-dose combination of Azilsartan and Amlodipine
  Arms: TAK-536CCB 20 mg/5 mg ＋Placebo (dual therapy)
Drug: TAK-536CCB + Hydrochlorothiazide — TAK-536CCB 20 mg/5 mg and Hydrochlorothiazide 6.25 mg tablets
  Other Names: Hydrochlorothiazide and fix-dose combination of Azilsartan and Amlodipine
  Arms: TAK-536CCB 20 mg/5 mg ＋HCTZ 6.25 mg (triple therapy)
Drug: Hydrochlorothiazide — TAK-536CCB placebo and Hydrochlorothiazide 6.25 mg tablets
  Arms: Placebo ＋HCTZ 6.25 mg (HCTZ monotherapy)
Drug: Hydrochlorothiazide — TAK-536CCB placebo and Hydrochlorothiazide 6.25 mg tablets x2
  Arms: Placebo ＋Hydrochlorothiazide 12.5 mg (HCTZ monotherapy)
Drug: TAK-536CCB + Hydrochlorothiazide — TAK-536CCB 20 mg/5 mg and Hydrochlorothiazide 6.25 mg tablets x2
  Other Names: Hydrochlorothiazide and fix-dose combination of Azilsartan and Amlodipine
  Arms: TAK-536CCB 20 mg/5 mg ＋HCTZ 12.5 mg (triple therapy)

SUMMARY:
The objective of this study is to compare the efficacy and safety of combined administration of TAK-536CCB (Fix-dose combination of Azilsartan and Amlodipine) and Hydrochlorothiazide (HCTZ) with those of TAK-536CCB in patients with Grade I or II essential hypertension.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, multicenter, phase 2/3 study to evaluate the efficacy and safety of combined administration of TAK-536CCB and Hydrochlorothiazide (HCTZ) with those of TAK-536CCB or Hydrochlorothiazide in patients with grade I or II essential hypertension.

This study consists of a 4-week single-blind placebo run-in period and a 10-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Grade I or II essential hypertension.
2. An office sitting systolic blood pressure of ≥ 150 and < 180 mmHg, and an office sitting diastolic blood pressure of ≥ 95 and < 110 mmHg during the placebo run-in period at Week -2 and Week 0.
3. Male or female aged 20 years or older at the time of providing informed consent.
4. Outpatient.

Exclusion Criteria:

1. Secondary hypertension, grade III hypertension or malignant hypertension.
2. An office sitting systolic blood pressure of ≥160 mmHg or sitting diastolic blood pressure of ≥100 mmHg recorded while on combined therapy with 3 or more antihypertensives within 4 weeks prior to the initiation of the placebo run-in period and at Week -4.

3 Evident white coat hypertension or white coat phenomenon. 4. Day-night reversed lifestyle, such as night-time workers. 5. Sleep apnea syndrome requiring treatment. 6. Have any of the cardiovascular disease or symptoms listed below:

* Heart disease: myocardial infarction (within 24 weeks before the placebo run-in period), coronary arterial revascularization (within 24 weeks before the placebo run-in period), severe valvular disease, atrial fibrillation, or following diseases which require medication: angina pectoris, congested heart failure, or arrhythmia.
* Cerebrovascular disease: cerebral infarction, cerebral hemorrhage (within 24 weeks before the placebo run-in period), or transient ischemic attack (within 24 weeks before the placebo run-in period).
* Vascular diseases: peripheral arterial disease with intermittent claudication, artery dissection, aneurysm
* Advanced hypertensive retinopathy: bleeding, exudation, or papilledema (within 24 weeks before the placebo run-in period).

  7. Clinically significant hepatic disorder. 8. Clinically significant renal impairment. 9. Significantly low or high Potassium or Sodium levels. 10. Complicated by gout, or had a past history of gout within 24 weeks prior to the initiation of the placebo run-in period, or complicated by hyperuricemia requiring medication.

  11. Diabetic subject on insulin treatment or poorly controlled type 2 diabetes mellitus.

  12. Have a malignant tumor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the office trough sitting diastolic blood pressure (DBP) | Baseline and Week 10
  Change in the office trough sitting DBP from the end of the placebo run-in period (baseline [Week 0]) to the end of the treatment period (Week 10, last observation carried forward [LOCF])

SECONDARY OUTCOMES:
Change from Baseline in the office trough sitting systolic blood pressure (SBP) | Baseline and Week 10
  Change in the office trough sitting SBP from the end of the placebo run-in period (baseline [Week 0]) to the end of the treatment period (Week 10, last observation carried forward [LOCF])
Proportion of patients achieving < 140/90 mmHg | 10 weeks
  Patients achieving < 140/90 mmHg refer to those meeting both of the following criteria:
  * A decrease to < 90 mmHg in office trough sitting DBP
  * A decrease to < 140 mmHg in office trough sitting SBP
Proportion of responders (140/90 mmHg criterion) | 10 weeks
  Patients who met either of the following conditions are regarded as responders (140/90 mmHg criterion).
  * A ≥ 20 mmHg decrease in office trough sitting SBP and a ≥ 10 mmHg decrease in the office trough sitting DBP
  * A decrease to < 140 mmHg in office trough sitting SBP and a decrease to < 90 mmHg in office trough sitting DBP
Frequency of adverse events( including vital sign, body weight, ECG findings and laboratory tests) | 10 weeks
  The frequency of adverse events by type, seriousness. Adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug to the last dose of study drug
Time profile of office trough sitting diastolic blood pressure | 10 weeks
Time profile of office trough sitting systolic blood pressure | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (13):
- Japan (13):
  - Touon-shi, Ehime
  - Fukuoka, Fukuoka
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Hanamaki-shi, Iwate
  - Morioka, Iwate
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Shinjuku-ku, Tokyo
  - Toyama, Toyama